CLINICAL TRIAL: NCT00876642
Title: Phase III Trial Comparing Best Supportive Care to Aloe Vera Gel as a Prophylactic Agent for Radiation Induced Skin Toxicity
Brief Title: Trial Comparing Best Supportive Care to Aloe Vera Gel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marilia Medicine School (Other)
Responsible Party: Gustavo Viani Arruda, Marilia Medicine school
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Oncoclinica-2009-02
Record Dates: First submitted 2009-04-05; First posted 2009-04-07 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Radiation Dermatitis
Keywords: Radiation dermatitis; best supportive care; Aloe vera gel; phase III study was to assess the effectiveness of aloe vera and vitamin E.
MeSH Terms: conditions — Radiodermatitis | interventions — Aloe vera gel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Aloe vera gel
- 2 (No Intervention)

INTERVENTIONS:
Drug: Aloe vera gel — The aloe vera gel which was commercially available, contained water, aloe vera, D-panthenol, triethanolamine, carbomer 934P, hyaluronic acid, potassium sorbate, diazolidinyl urea, methylparaben, and propylparaben.
  Arms: 1

SUMMARY:
Radiation therapy (RT) has been a component of breast cancer treatment for almost 100 years. Although initially used for the treatment of chest wall recurrences after mastectomy and for advanced inoperable disease, RT has evolved into a critical component of early therapy for women with an intact breast following lumpectomy and for mastectomized women who are at high risk for local failure. Currently breast cancer patients need a multidisciplinary management including surgery, chemotherapy and radiotherapy, radiotherapy has a significant role in loco regional control of the disease. It is estimated that 87% of these women will develop some degree of radiation-induced dermatitis, varying from mild to brisk erythema or even moist desquamation.

Topical agents, such as corticosteroid creams and other products including Aquaphor (Beirsdorf Inc, Wilton, CT), and trolamine (Biafine; Genmedix Ltd, France), are commonly prescribed at the onset of radiation dermatitis or, in some institutions, at the beginning of radiotherapy.

The aim of this randomized phase III study was to assess the effectiveness of aloe vera cream for the prevention of acute radiation-induced dermatitis of grade 2 or higher during postoperative radiotherapy for breast cancer, compared to best supportive care. The secondary objectives were to assess pain, treatment interruption as a result of skin reactions, and the quantity of life during the treatment.

ELIGIBILITY:
Inclusion Criteria:

* The women had to be 18 to 75 years of age with a nonmetastatic breast adenocarcinoma treated by either lumpectomy or mastectomy with or without adjuvant postoperative chemotherapy or hormonal treatment, and referred to the Department of Radiotherapy for postoperative radiotherapy. Concomitant chemotherapy was allowed.

Exclusion Criteria:

* Women with bilateral cancer, patients who were allergic to either of the two agents, and pregnant women were excluded.
* No rash, ulceration, bleeding, or unhealed scar was allowed in the treatment area.
* Patients were excluded for: prior radiation therapy (RT), mastectomy, skin involvement by tumor, history of, or current connective tissue disorder, medical contraindication (allergy or sensitivity) to Aloevera or planned BSC, and inability to comply with treatment regime. The use of bolus was prohibited.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Acute radiation-induced dermatitis of grade 2 or higher during postoperative radiotherapy for breast cancer.

SECONDARY OUTCOMES:
quality of life,interruptions of treatment and pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustavo Viani, Marília, Sao Paulo\brazil, Brazil